CLINICAL TRIAL: NCT03455036
Title: The Mysterious on/Off Itch and Erythema During Whole Body Vibration Exercise
Acronym: VIBRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-02009
Record Dates: First submitted 2018-02-27; First posted 2018-03-06 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Itch; Athlete
Keywords: whole body vibration, erythema, tryptase, unpleasantness
MeSH Terms: conditions — Pruritus; Erythema

STUDY DESIGN:
Intervention Model Description: The design of the study is a single-centre cross-sectional single-arm intervention study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole body vibration training (Experimental): Healthy female subjects complete whole body vibration training (10 x 1 min exposure)
  Interventions: Other: Whole body vibration training

INTERVENTIONS:
Other: Whole body vibration training — 10 x 1 min whole body vibration exposure

SUMMARY:
Intense itch on the legs sometimes associated with redness can be adverse effects of whole body vibration (WBV) according to own observations and numerous posts in non-professional online-blogs. To the investigators' knowledge, the appearance of itch and/or a rash during WBV exercise has not yet been described.

The research objectives are:

1. To determine the effect of WBV on itch rating and its unpleasantness and on skin changes.
2. To determine the effect of WBV on immunoglobulin E (IgE) and serum tryptase

DETAILED DESCRIPTION:
Objectives Intense itch on the legs sometimes associated with redness can be adverse effects of WBV according to the investigators observations and numerous posts in non-professional online-blogs. To the investigators knowledge, the appearance of itch and/or a rash during WBV exercise has not yet been described.

The objectives of this study are:

1. to determine the effect of WBV on itch rating and its unpleasantness and on skin changes.
2. to determine the effect of WBV on serum tryptase.

Hypothesis The working hypothesis is that repeated WBV leads to an increase of itching and erythema. Further investigators hypothesize that repeated WBV does not lead to an increase in serum tryptase.

Inclusion and exclusion criteria will be evaluated. Subjects will be instructed to not shave their legs one week before the intervention day and to shave only the left leg from the ankle to the knee on the day prior to the intervention day.

On the intervention day, subjects will be informed in detail about the study protocol and written informed consent will be collected. If a pregnancy cannot be excluded (days from last menstruation) subjects are instructed to do a pregnancy test. Then, a blood sample will be taken. Subsequently, subjects will be instructed to stand on the vibration plate (Galileo 900) in a slightly crouched position with their hands loosely resting on the rail. Subjects will complete ten 1-minute WBV repetitions interspaced by 1-minute breaks in seated position. During each break, subjects will rate the itch intensity, and skin changes will be captured. Sixty minutes after the last WBV repetition, another blood sample will be taken. Subjects will rest until itch and erythema return to baseline. During resting phase subjects will fill in the Eppendorf itch questionnaire and the Erlanger atopy score.

ELIGIBILITY:
Inclusion Criteria:

* age 18-35 years
* female
* Informed Consent as documented by signature (Appendix Informed Consent Form)

Exclusion Criteria:

* itchy skin diseases
* hay fever
* asthma
* chronic venous insufficiency
* peripheral artery disease
* musculoskeletal diseases or injuries affecting the legs, hips and pelvis
* BMI < 17 and > 35 kg/m2
* pregnancy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female participants only
Enrollment: 20 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Itch intensity | 0 months
  0 to 10 numerical rating scale (NRS) (best score: 0 - no itch; worst score: 10)

SECONDARY OUTCOMES:
Erlanger atopy score | 0 months
  Erlanger atopy score (best score: 0 - no atopy; worst score: 100)
Itch characteristics | 0 months
  measured using Eppendorf itch questionnaire
Itch unpleasantness | 0 months
  0 to 10 numerical rating scale (NRS) (best score: 0 - no unpleasantness; worst score: 10)
Skin surface temperature | 0 months
  assessed using a infrared thermal camera
Erythema intensity | 0 months
  assessed using an erythema meter
Total immunoglobulin E (IgE) concentration | 0 months
  Serum
Tryptase concentration | 0 months
  serum

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Muendermann, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No